CLINICAL TRIAL: NCT05590247
Title: Role of Intermittent Fasting on Disease Severity and Quality of Life in Psoriasis and Psoriatic Arthritis
Brief Title: Role of Intermittent Fasting in Psoriasis and Psoriatic Arthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Psoriasis Foundation (Other)
Responsible Party: Principal Investigator, Ben H Kaffenberger, Dr., Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022H0186
Record Dates: First submitted 2022-10-05; First posted 2022-10-21 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Psoriasis; Psoriatic Arthritis
Keywords: fasting; intermittent
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic; Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-blind parallel group randomized control trial. Participants will be identified through an electronic medical record search for established patients within the Ohio State Dermatology practice with a diagnosis of mild-to-moderate psoriasis. Patients will then be asked to join the study and subsequently given information to consent. Patients in the control group will be offered entry into the intermittent fasting group after the commencement of the study as an incentive to participate.
Who Masked: Care Provider, Investigator
Masking Description: Care provider and investigator are blinded to the arm, but patient has to know which diet to follow and outcomes assessor assigned the groups and has to counsel patients accordingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermittent Fasting Group (Experimental): Patients in this group will do intermittent fasting dieting for 12 weeks, meaning they will only eat for 8 hours per day. They may choose whichever 8 hours they want. Only water can be consumed during the fasting period. For the last 12 weeks of the study, they will resume their normal diet.
  Interventions: Behavioral: Intermittent Fasting Diet
- Standard Routine Diet Group (No Intervention): Patients will continue with their normal diets for the 24 week duration of the study.

INTERVENTIONS:
Behavioral: Intermittent Fasting Diet — Patients will follow the 16: 8 traditional intermittent fasting model, where they may only consume calories during 1 continuous 8-hour period of the day. Water may be consumed during fasting.
  Other Names: fasting; intermittent energy restriction
  Arms: Intermittent Fasting Group

SUMMARY:
Our study aims to determine whether intermittent fasting (IMF) is a valid method to improve psoriasis and psoriatic arthritis (PsA) disease severity and quality of life. Patients within OSU Dermatology with psoriasis and/or psoriatic arthritis will be enrolled in a dietary intervention for a 24-week period. A prospective, single-blind parallel group randomized control trial will include an IMF dietary intervention group and a standard routine diet group for a duration of 24 weeks. After the initial 12 weeks of the dietary intervention, patients will be followed for an additional 12 weeks to assess changes in their disease state and quality of life after returning to their initial dietary routines. In total, the study will be 24 weeks. Baseline assessment will consist of standard psoriasis and PsA clinical parameters; evaluation will be performed by a blinded physician. These parameters will be reassessed every 4 weeks via video visit for the three month duration of the study, and then again at the 24-week conclusion of the study. In addition, each visit will assess patient-reported outcomes using dermatology-specific quality of life indices. Biometric measurements of weight, height, BMI, and waist-to-hip ratio will be recorded at baseline and all subsequent visits. Dietary adherence will be assessed by virtual check-in visits, and dietary guidance will be provided and reviewed at each visit by the research coordinator. A physician or the research coordinator will be available for questions between times of data collection. The primary outcome measure will be feasibility of a larger study, which will be determined at the initial 12-week timepoint. This data is vital to determine effect size and dropout frequency for future studies. Secondary outcomes will include changes in clinical indices, biometric measurements, and quality of life indices at 12 weeks after randomization and at the end of the 24-week study. Achievement of a 5% weight reduction at 12 weeks, and a 10-15% weight reduction at 24 weeks will be additional secondary endpoints. Data for each patient will be stored in a password-protected and encrypted REDCAP database on a secure OSU server.

DETAILED DESCRIPTION:
Aim 1: Assess the feasibility of a larger study testing the association between intermittent fasting and disease severity in patients with psoriasis using psoriasis-specific clinical indices and patient-reported psoriasis outcomes.

The investigators will conduct a prospective, single-blind parallel group randomized control trial. Participants will be identified through an electronic medical record search for established patients within the Ohio State Dermatology practice with a diagnosis of mild-to-moderate psoriasis. Patients will then be asked to join the study and subsequently given information to consent. Patients in the control group will be offered entry into the intermittent fasting group after the commencement of the study as an incentive to participate.

Setting: The clinical setting will be the outpatient dermatology clinic sites for the Ohio State University Wexner Medical Center, Columbus, OH. The sites have access to measurement equipment, well-lit examination rooms, clinical trial support, and convenient locations for patient access.

Study Procedures: Patients will receive information regarding their dietary modifications before the start of the study; they will also be randomized to their group at this time. In the IMF group of the study, subjects will be permitted to eat food of any type and quantity for 8 hours of each day at any timing. Patients in the standard routine dietary guidance group are encouraged to continue their current diet while recording their first and last meal of the day until the first data collection. By doing this, the investigators will ensure that there is a difference in total energy consumption time between the IMF group and our controls. After the first 12 weeks of the study and subsequent data collection, patients will be permitted to resume their normal dietary habits for the remaining 12 weeks of the study.

Random Allocation: Following consent, the participants who meet the inclusion criteria will be block randomized by presence of PsA and time in a 1:1 ratio to either the IMF diet intervention or standard routine dietary guidance. Recruitment will ensure at least 20% of each group contains patients with PsA. The assessing physician investigator will be blinded to the group assignment of each patient, although the research coordinator will not be blinded. Patients cannot reasonably be blinded to their assignment. Data for each patient will be stored in a password-protected and encrypted REDCAP database on a secure OSU server. Each patient will receive a random numerical identity in the database which their data points will be associated with. Data access is role-based and limited to PI, research coordinator, statistician, and support staff.

Early stopping rules: Early stop permitted due to illness or lack of adherence; data will be included under the intention-to-treat (ITT) assumption.

Monitoring Plan: Safety monitoring will be patient-reported when patients come to clinical site and in between checkpoints if needed. Due to COVID-19, adjustments for electronic visitations will be allowable if patients can appropriately document all areas of involvement as well as take updated biometric measurements.

Aim 2: Assess the feasibility of a larger study testing the association between intermittent fasting and disease severity in patients with psoriatic arthritis using standardized DAPSA score and patient-reported outcomes

Setting: As in Aim 1, the clinical setting will be the outpatient dermatology clinic sites for the Ohio State University Wexner Medical Center, Columbus, OH. The resources and personnel at these sites are also appropriate for this aim. Design: In this aim, data points to be collected will be the DAPSA score, as well as scoring systems for enthesitis and dactylitis. Quality of life will be assessed using HRQL score.

Study Procedures: After the patient has consented, the patient will be block randomized as in Aim 1. Initial baseline assessment will be performed by a blinded physician. Baseline assessment will consist of DAPSA, enthesitis, and dactylitis indices. Health-related quality of life (HRQL) survey will be administered to patients at baseline and 12 and 24-week timepoints. All other items that are collected in Aim 1 will also be collected in this group.

All other aspects of Aim 2 not mentioned in this section are the same as in Aim 1.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Established patient at the clinical site with a diagnosis of mild to moderate plaque psoriasis despite treatment
* Ability to consent and follow dietary instructions
* Overweight (BMI ≥ 25)
* No change in systemic psoriasis treatment for 6 weeks

Exclusion Criteria:

* Pregnancy and/or breastfeeding
* Insulin-dependent diabetics
* Severe heart, kidney, and liver disease
* Obesity due to medical condition
* Use of medical treatment for weight reduction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Disease activity (skin) by PASI scoring | 0 weeks (baseline), 12 weeks, 24 weeks
  Measured by Psoriasis Area Severity Index (PASI; scored 0-72, 72 is worst).
  *Note: calculated for both psoriasis and psoriatic arthritis patients.
  This score is a calculation based on assessment of erythema, desquamation, and induration in four distinct body areas: head/neck, trunk, upper extremities, and lower extremities.
Change in Disease activity (joints) by PsARC scoring | 0 weeks (baseline), 12 weeks, 24 weeks
  PsARC (Psoriatic Arthritis Response Criteria)
  *Note: only for psoriatic arthritis patients
  Response is defined by improvement in at least 2 of the 4 following measures, one of which must be joint swelling or tenderness, and no worsening in any of the 4 measures:
  1. Patient generalized assessment (PGA) of articular disease (0-4, 4 being most severe)
  2. Investigator generalized assessment (IGA) of articular disease (0-4, 4 being most severe)
     *for 1-2: improvement = decrease by one category, worsening = increase by one category.
  3. Joint pain/tenderness score (numeric sum of number of involved joints)
  4. Joint swelling score (numeric sum of number of involved joints) *for 3-4: improvement = decrease by 30%, worsening = increase by 30%.

SECONDARY OUTCOMES:
Patient Quality of life (Patient experience with their disease) by DLQI scoring | 0 weeks (baseline), 12 weeks, 24 weeks
  Psoriasis: quality of life assessed via Dermatology Life Quality Index (DLQI; scored 0-30, 30 is worst). Psoriatic arthritis: quality of life assessed via Health-related Quality of Life Index (HRQL).
  *Note: patients with psoriatic arthritis will complete both surveys.
Amount of skin involvement | 0 weeks (baseline), 12 weeks, 24 weeks
  Body surface area (0-100%)
Disease activity (overall) | 0 weeks (baseline), 12 weeks, 24 weeks
  Physician's Global Assessment (score 0-4, 4 being worst)
Enthesitis and Dactylitis Assessment | 0 weeks (baseline), 12 weeks, 24 weeks
  Will be scored on presence/absence of dactylitis and enthesitis based on physical exam.
Disease activity (nails) | 0 weeks (baseline), 12 weeks, 24 weeks
  Nail Psoriasis Severity Index (NAPSI; 0-160, 160 is worst) The nail is divided into quadrants, and each nail is given a score for nail bed psoriasis (0-4) and nail matrix psoriasis (0-4) depending on the presence of the following features of nail psoriasis in that quadrant.
  1. Evaluation 1: Nail matrix. In each quadrant of the nail, nail matrix psoriasis is evaluated by presence of any of the nail matrix features (pitting, leukonychia red spots in the lunula, crumbling): 0 for none, 1 if present in 1quadrant of the nail, 2 if present in 2 quadrants of the nail, 3 if present in 3 quadrants of the nail, and 4 if present in 4 quadrants of the nail.
  2. Evaluation 2: Nail bed. Nail bed psoriasis is evaluated by the presence of any of the nail bed features (onycholysis, splinter hemorrhages, subungual hyperkeratosis, "oil drop" (salmon patch dyschroma): 0 for none, 1 for 1 quadrant only, 2 for 2 quadrants,3 for 3 quadrants, and 4 for 4 quadrants.
  3. Each nail gets a matrix score and
Weight | 0 weeks (baseline), 12 weeks, 24 weeks
  Weight will be obtained in kilograms using traditional clinical scale.
Height | 0 weeks (baseline), 12 weeks, 24 weeks
  Height will be obtained in meters using traditional clinical scale.
Body Mass Index (BMI) | 0 weeks (baseline), 12 weeks, 24 weeks
  BMI assessed by obtaining weight (kg) and height (m) from traditional clinical scale and calculating.
Waist-to-hip ratio | 0 weeks (baseline), 12 weeks, 24 weeks
  Waist-to-hip ratio will be measured using tape measure in centimeters and reported as a ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin H Kaffenberger, MD, MS, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Damiani G, Watad A, Bridgewood C, Pigatto PDM, Pacifico A, Malagoli P, Bragazzi NL, Adawi M. The Impact of Ramadan Fasting on the Reduction of PASI Score, in Moderate-To-Severe Psoriatic Patients: A Real-Life Multicenter Study. Nutrients. 2019 Jan 27;11(2):277. doi: 10.3390/nu11020277. PMID 30691245
- [Background] Ford AR, Siegel M, Bagel J, Cordoro KM, Garg A, Gottlieb A, Green LJ, Gudjonsson JE, Koo J, Lebwohl M, Liao W, Mandelin AM 2nd, Markenson JA, Mehta N, Merola JF, Prussick R, Ryan C, Schwartzman S, Siegel EL, Van Voorhees AS, Wu JJ, Armstrong AW. Dietary Recommendations for Adults With Psoriasis or Psoriatic Arthritis From the Medical Board of the National Psoriasis Foundation: A Systematic Review. JAMA Dermatol. 2018 Aug 1;154(8):934-950. doi: 10.1001/jamadermatol.2018.1412. PMID 29926091
- [Background] Di Minno MN, Peluso R, Iervolino S, Russolillo A, Lupoli R, Scarpa R; CaRRDs Study Group. Weight loss and achievement of minimal disease activity in patients with psoriatic arthritis starting treatment with tumour necrosis factor alpha blockers. Ann Rheum Dis. 2014 Jun;73(6):1157-62. doi: 10.1136/annrheumdis-2012-202812. Epub 2013 Jun 14. PMID 23771989
- [Background] Adawi M, Damiani G, Bragazzi NL, Bridgewood C, Pacifico A, Conic RRZ, Morrone A, Malagoli P, Pigatto PDM, Amital H, McGonagle D, Watad A. The Impact of Intermittent Fasting (Ramadan Fasting) on Psoriatic Arthritis Disease Activity, Enthesitis, and Dactylitis: A Multicentre Study. Nutrients. 2019 Mar 12;11(3):601. doi: 10.3390/nu11030601. PMID 30871045
- [Background] Takeshita J, Grewal S, Langan SM, Mehta NN, Ogdie A, Van Voorhees AS, Gelfand JM. Psoriasis and comorbid diseases: Epidemiology. J Am Acad Dermatol. 2017 Mar;76(3):377-390. doi: 10.1016/j.jaad.2016.07.064. PMID 28212759
- [Background] Afifi L, Danesh MJ, Lee KM, Beroukhim K, Farahnik B, Ahn RS, Yan D, Singh RK, Nakamura M, Koo J, Liao W. Dietary Behaviors in Psoriasis: Patient-Reported Outcomes from a U.S. National Survey. Dermatol Ther (Heidelb). 2017 Jun;7(2):227-242. doi: 10.1007/s13555-017-0183-4. Epub 2017 May 19. PMID 28526915
- [Background] Pona A, Haidari W, Kolli SS, Feldman SR. Diet and psoriasis. Dermatol Online J. 2019 Feb 15;25(2):13030/qt1p37435s. PMID 30865402
- [Background] Fernandez-Armenteros JM, Gomez-Arbones X, Buti-Soler M, Betriu-Bars A, Sanmartin-Novell V, Ortega-Bravo M, Martinez-Alonso M, Gari E, Portero-Otin M, Santamaria-Babi L, Casanova-Seuma JM. Psoriasis, metabolic syndrome and cardiovascular risk factors. A population-based study. J Eur Acad Dermatol Venereol. 2019 Jan;33(1):128-135. doi: 10.1111/jdv.15159. Epub 2018 Jul 17. PMID 29953676
- [Background] Shelling ML, Kirsner RS. Practice gaps. Gaining insights into the relationship of obesity, weight loss, and psoriasis. JAMA Dermatol. 2013 Jul;149(7):801-2. doi: 10.1001/jamadermatol.2013.3383. No abstract available. PMID 23752561
- [Background] Debbaneh M, Millsop JW, Bhatia BK, Koo J, Liao W. Diet and psoriasis, part I: Impact of weight loss interventions. J Am Acad Dermatol. 2014 Jul;71(1):133-40. doi: 10.1016/j.jaad.2014.02.012. Epub 2014 Apr 4. PMID 24709272
- [Background] Zuccotti E, Oliveri M, Girometta C, Ratto D, Di Iorio C, Occhinegro A, Rossi P. Nutritional strategies for psoriasis: current scientific evidence in clinical trials. Eur Rev Med Pharmacol Sci. 2018 Dec;22(23):8537-8551. doi: 10.26355/eurrev_201812_16554. PMID 30556896
- [Background] Wu AG, Weinberg JM. The impact of diet on psoriasis. Cutis. 2019 Aug;104(2S):7-10. PMID 31634384
- [Background] de Cabo R, Mattson MP. Effects of Intermittent Fasting on Health, Aging, and Disease. N Engl J Med. 2019 Dec 26;381(26):2541-2551. doi: 10.1056/NEJMra1905136. No abstract available. PMID 31881139
- [Background] Mattson MP, Longo VD, Harvie M. Impact of intermittent fasting on health and disease processes. Ageing Res Rev. 2017 Oct;39:46-58. doi: 10.1016/j.arr.2016.10.005. Epub 2016 Oct 31. PMID 27810402
- [Background] Anton SD, Moehl K, Donahoo WT, Marosi K, Lee SA, Mainous AG 3rd, Leeuwenburgh C, Mattson MP. Flipping the Metabolic Switch: Understanding and Applying the Health Benefits of Fasting. Obesity (Silver Spring). 2018 Feb;26(2):254-268. doi: 10.1002/oby.22065. Epub 2017 Oct 31. PMID 29086496
- [Background] Yang F, Liu C, Liu X, Pan X, Li X, Tian L, Sun J, Yang S, Zhao R, An N, Yang X, Gao Y, Xing Y. Effect of Epidemic Intermittent Fasting on Cardiometabolic Risk Factors: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Front Nutr. 2021 Oct 18;8:669325. doi: 10.3389/fnut.2021.669325. eCollection 2021. PMID 34733872
- [Background] Jensen P, Zachariae C, Christensen R, Geiker NR, Schaadt BK, Stender S, Hansen PR, Astrup A, Skov L. Effect of weight loss on the severity of psoriasis: a randomized clinical study. JAMA Dermatol. 2013 Jul;149(7):795-801. doi: 10.1001/jamadermatol.2013.722. PMID 23752669
- [Background] Bragazzi NL, Sellami M, Salem I, Conic R, Kimak M, Pigatto PDM, Damiani G. Fasting and Its Impact on Skin Anatomy, Physiology, and Physiopathology: A Comprehensive Review of the Literature. Nutrients. 2019 Jan 23;11(2):249. doi: 10.3390/nu11020249. PMID 30678053
- [Background] Rynders CA, Thomas EA, Zaman A, Pan Z, Catenacci VA, Melanson EL. Effectiveness of Intermittent Fasting and Time-Restricted Feeding Compared to Continuous Energy Restriction for Weight Loss. Nutrients. 2019 Oct 14;11(10):2442. doi: 10.3390/nu11102442. PMID 31614992
- [Background] Plikus MV, Van Spyk EN, Pham K, Geyfman M, Kumar V, Takahashi JS, Andersen B. The circadian clock in skin: implications for adult stem cells, tissue regeneration, cancer, aging, and immunity. J Biol Rhythms. 2015 Jun;30(3):163-82. doi: 10.1177/0748730414563537. Epub 2015 Jan 13. PMID 25589491
- [Background] Adawi M, Watad A, Brown S, Aazza K, Aazza H, Zouhir M, Sharif K, Ghanayem K, Farah R, Mahagna H, Fiordoro S, Sukkar SG, Bragazzi NL, Mahroum N. Ramadan Fasting Exerts Immunomodulatory Effects: Insights from a Systematic Review. Front Immunol. 2017 Nov 27;8:1144. doi: 10.3389/fimmu.2017.01144. eCollection 2017. PMID 29230208
- [Background] Macklis P, Adams KM, Li D, Krispinsky A, Bechtel M, Trinidad J, Kaffenberger J, Kumar P, Kaffenberger BH. The impacts of oral health symptoms, hygiene, and diet on the development and severity of psoriasis. Dermatol Online J. 2019 Jul 15;25(7):13030/qt85z4t7hq. PMID 31450285
- [Background] Macklis PC, Tyler K, Kaffenberger J, Kwatra S, Kaffenberger BH. Lifestyle modifications associated with symptom improvement in hidradenitis suppurativa patients. Arch Dermatol Res. 2022 Apr;314(3):293-300. doi: 10.1007/s00403-021-02233-y. Epub 2021 Apr 23. PMID 33893517